CLINICAL TRIAL: NCT03342885
Title: The Effect of Sleep Ergonomics on Pain Low Back Pain
Brief Title: Sleep Ergonomics in Low Back Pain
Acronym: SLEEPLBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Finland Hospital District (Other)
Responsible Party: Principal Investigator, Jari Ylinen, Chief Physician, Central Finland Hospital District
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnro1E/2017
Record Dates: First submitted 2017-10-30; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Sleep ergonomics
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants enrolled into the intervention group receive specific sleep ergonomics guidance
  Interventions: Behavioral: Specific sleep ergonomics guidance
- Control group (Active Comparator): Participants enrolled into the control group will receive general sleep ergonomics guidance
  Interventions: Behavioral: General sleep ergonomics guidance

INTERVENTIONS:
Behavioral: Specific sleep ergonomics guidance — Participants receive a detailed instruction in sleep ergonomics. Participants are instructed to maintain either side lying or supine sleeping posture, depending on which is less painful. Neutral position of spine supported by specific placement of body pillow. Changing of posture during sleep is prevented. The participants are recommended to replace their mattress if they feel that it is too hard or too soft. Instruction is given by a physiotherapist during one personal therapy session and the participants also receive a printed instruction.
  Arms: Intervention group
Behavioral: General sleep ergonomics guidance — Participants are instructed find most comfortable sleeping posture by personal preference and to avoid painful posture. The participants are recommended to replace their mattress if they feel that it is too hard or too soft. Instruction is given by a physiotherapist during one personal therapy session and the participants also receive a printed instruction.
  Arms: Control group

SUMMARY:
The aim of this study is to investigate the effect of sleep ergonomics guidance given by physiotherapist on pain and disability in patients with low back pain. In this randomized controlled trial participants are assigned either into the intervention or the control group. The intervention group will receive detailed instruction on sleeping ergonomics whereas the control group will only be instructed to avoid painful sleeping posture. The initial hypothesis is that in the intervention group pain and disability will decrease more compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Low Back Pain
* Pain during sleep or

Exclusion Criteria:

* Fibromyalgia
* Inflammatory rheumatic disease
* Severe depression or other psychiatric diagnosis
* Previously received specific guidance in sleep ergonomics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Visual Analog Scale (VAS) | Change from baseline to 12 month follow-up
  Low back pain reported with Visual Analog Scale (VAS) during rest, after getting up and during day; 0-100 mm scales, 0 mm = no pain, 100 mm = worst possible pain. Change from baseline to 12 month follow-up is reported in mm for each sub-scale (during rest, after getting up and during day).
Oswestry Disability Index (ODI) score | Change from baseline to 12 month follow-up
  Oswestry Disability Index Finnish version 2.0 total score (scale 0-100%): 0 = minimal disability, 100 = bed-bound or exaggeration of symptoms; and sub-scores (scale 0-5): 0 = minimal disability, 5 = worst disability. Change is reported for total ODI score and sub-scores from baseline to 12 month follow-up.

SECONDARY OUTCOMES:
Reported amount of sleep | Change from baseline to 12 month follow-up
  Perceived sufficiency of sleep based on question: "Do you feel that you have got sufficient sleep during last week?", reported with 5 step Likert scale (scale 1-5), 1 = not sufficient at all, 5 = totally sufficient. Change in perceived sufficiency of sleep is reported from baseline to 12 month follow-up.
Number of sick leave days | Change from baseline to 12 month follow-up
  Number of sick leave days during last 12 months as reported by the participant. Change in sick leave days during last 12 months is reported from baseline to 12 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jari Ylinen, MD, Principal Investigator — Central Finland Hospital District
Locations (1):
- Central Finland Central Hospital, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: No